CLINICAL TRIAL: NCT02648100
Title: Identification and Treatments of Basal Like Bladder Cancer (Study on Human Tumor Samples and Animal Models)
Brief Title: Basal Like Bladder Cancer : Signature and Therapeutic
Acronym: DIATRIBBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Paris 12 Val de Marne University (Other); Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: NI 13021
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Muscle Invasive Bladder Cancer; Molecular Taxonomy
Keywords: Muscle invasive bladder cancer; Basal subtype; Anti-EGFR treatment; Nanostring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor tissue : frozen (n=120), FFPE (n=911)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: 120 patients from Carte d'Identité des Tumeurs (CIT), Henri Mondor and Foch hospitals.
  Interventions: Other: biomarker study
- B: 510 cystectomy patients operated between 2005 and 2010 in Henri Mondor and Foch hospitals.
  Interventions: Other: biomarker study
- C: 188 patients treated by cystectomy and adjuvant chemotherapy for locally advanced bladder cancer from a national multicentric study.
  Interventions: Other: biomarker study
- D: 93 patients from the clinical trial GETUG 19 (UNICANCER)
  Interventions: Other: biomarker study

INTERVENTIONS:
Other: biomarker study

SUMMARY:
Muscle invasive (MIBC) and/or metastatic bladder cancer is associated with poor prognosis and no target therapies for this pathology are currently validated. By 40 gene expression signature realized on frozen samples, we have previously identified an aggressive sub-class of MIBC, called basal. This sub-class (20% of MIBC) showed strong EGFR dependence in vitro and in vivo (Rebouissou et al. Science Translational Medicine 2014). This observation suggests a possible response to EGFR targeted therapy in patients of this subgroup. Our aim is to establish a standard diagnostic tool to differentiate the basal subtype of bladder cancer and evaluate the effect of anti-EGFR therapy, by analyzing previous clinical trial (GETUG19) and preclinical models, which compare the classical chemotherapy to anti-EGFR associated chemotherapy.

DETAILED DESCRIPTION:
The aim of this study is:

1. To validate a diagnostic test for formalin-fixed paraffin-embedded (FFPE) samples by Nanostring technology, using the 40 genes signature as reference. First, we will compare frozen and FFPE tissues (n=120), to establish a transcriptional signature in FFPE samples. Secondly, to further characterize basal subtype of bladder cancer, we will study the mutational and gain/loss landscape and immunohistochemistry markers in a new series of tumors after classifying them by our gene signature (n=510). These characteristics will be included in a new signature by defining the optimal prediction discrimination AIC et Net Reclassification Index.
2. To assess the prognosis after cisplatine treatment in 510 patients treated by cystectomy with or without adjuvant chemotherapy (pT2/pT3/pT4, N0 or N+) and in another multicentric series of 188 patients treated by cystectomy and adjuvant chemotherapy (pT3/pT4 et/ou N+). Uni and multi variant analysis will be realized by adjusted Cox model, and the added value of basal subtype as compared to standard prognostic factors will be evaluated. The propensity score will be realized to assess the association of basal subtype and response to chemotherapy. The anti-EGFR response will be analyzed in the clinical trial GETUG19 which uses Panitumumab in patients with metastatic urothelial carcinomas (n=93)
3. To study the treatment response in preclinical models. We characterized previously preclinical murine models derived from xenografts of MIBC (n=14 and new xenografts will be added). We will study the effect of anti-EGFR alone or in combination with chemotherapy in basal and non basal subtypes of xenografts.

By this study we will be able to better characterize the basal subtype of bladder cancer and confirm its aggressive behaviour as compared to other subtypes of MIBC. These results will further help to establish new clinical trials which include anti-EGFR in patients of basal subtype.

ELIGIBILITY:
Inclusion Criteria:

Muscle invasive bladder cancer Treatment by cystectomy Adjuvant chemotherapy for 3rd cohort Clinical trial GETUG 19 for 4th cohort

Exclusion Criteria:

FFPE material not available Follow-up data not available

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Bladder Cancer from 4 cohorts
  * 2 observational cohorts of patients with muscle invasive bladder cancer (all stages) from two Henri Mondor (Créteil) and Foch (Suresnes) hospitals
  * 1 multicentric observational cohort of patients with locally advanced muscle invasive bladder cancer trated by adjuvantchemotherapy after cystectomy
  * 1 clinical trial GETUG 19 (MVAC + panitumumab)
Sampling Method: Non-Probability Sample
Enrollment: 911 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Specific survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yves ALLORY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Yes